CLINICAL TRIAL: NCT04984330
Title: Selinexor for Treatment of Light Chain Amyloidosis With Relapsed/Refractory Disease
Acronym: STARR
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-01023225
Record Dates: First submitted 2021-07-29; First posted 2021-07-30 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Amyloid; Amyloidosis; AL Amyloidosis
MeSH Terms: conditions — Alzheimer Disease; Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — selinexor; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- selinexor/ dexamethasone (Sd) (Experimental): Selinexor • 60mg PO once weekly on days 1, 8, 15, 22 until disease progression or toxicity
  Dexamethasone
  • 20 mg PO administered 30-60 minutes prior to selinexor on days 1, 2, 8, 9, 15, 16, 22, 23
  Interventions: Drug: Selinexor; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — Selinexor will be given orally at a dose of 60mg once weekly on the first day of the week (day 1, 8, 15, and 22) for Cycle 1 and up to Cycle 12.
Drug: Dexamethasone — Dexamethasone will be given orally at a dose of 20mg, if tolerated, or at a reduced dose if required, 30 to 60 minutes prior to selinexor for first 2 days of each week only (days 1, 2, 8, 9, 15, 16, 22, and 23 of each cycle).

SUMMARY:
The purpose of this study is to test the safety and efficacy of Selinexor and Dexamethasone and see what effects it has on AL amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary AL amyloidosis
* Relapsed and/or refractory AL amyloidosis
* Measurable disease
* Male or female patients 18 years or older
* Able to give voluntary written consent
* Eastern Cooperative Oncology Group performance status and/or other performance status 0, 1, or 2.
* Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3.
* Total bilirubin ≤ 1.5 × the upper limit of the normal range (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN.
* Calculated creatinine clearance ≥ 30 mL/min

Exclusion Criteria:

* Non-AL amyloidosis
* Clinically overt myeloma
* Prior exposure to Selinexor
* Clinically significant cardiac disease
* Severe obstructive airway disease
* Female patients who are lactating or have a positive serum pregnancy test during the screening period
* Planned high-dose chemotherapy and autologous stem cell transplantation within 6, 28-day treatment cycles after starting on treatment
* Failure to have fully recovered (ie, ≤ Grade 1 toxicity) from the reversible effects of prior chemotherapy.
* Major surgery within 14 days before enrollment.
* Radiotherapy within 14 days before enrollment.
* Infection requiring systemic intravenous antibiotic therapy or other serious infection within 14 days before study enrollment. Systemic treatment, within 14 days before the first dose, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, see Appendix 11.7), or use of Ginkgo biloba or St. John's wort.
* Positive for human immunodeficiency virus (HIV), hepatitis B, and hepatitis C
* Serious medical or psychiatric illness
* GI disease or GI procedure that could interfere with the oral absorption or tolerance including difficulty swallowing
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Participation in another clinical trials involving investigational agents within 30 days of starting this trial
* Peripheral neuropathy (grade 2 with pain or grade 3 or higher).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Compare number of dose limiting toxicity (DLT) occurence to measure safety and toxicity | approximately 12 months
  Safety and toxicity will be determined by how many occurrence of dose limiting toxicity (DLT) occured during 12 months of treatment for each subject

SECONDARY OUTCOMES:
Compare Hematologic Overall Response Rate (ORR) | approximately 12 months
  Comparing proportion of subjects with Complete Response (CR), Very Good Partial Response (VGPR), Partial Response (PR), No Response (NR) and Progressive Disease (PD)
Hematologic Very Good Partial Response (VGPR) or better rate | approximately 12 months
  Percentage of subjects that achieved Very Good Partial Response (VGPR) or better response
Hematologic Complete Response (CR) rate | approximately 12 months
  Percentage of subjects that achieved Complete Response (CR)
Stringent dFLC response rate | approximately 12 months
  Percentage of subjects that has stringent dFLC (dFLC is defined as the difference in involved amyloidogenic and uninvolved serum-free light chains).
Number of patients with peripheral blood mass spectrometry for monoclonal protein detection (MALDI-TOF) | End of Study (approximately 3 years)
  For each subject, detection of monoclonal protein will be analyzed at screening, day 1 of each cycle (only when in ≥VGPR), at each end of treatment (EOT) visits, and day 1 of each post-treatment follow, up until PD or 24 months, whichever occurs first.
minimal residual disease (MRD) negative CR/VGPR rate | approximately 12 months
  Percentage of subjects that is MRD negative when in complete response (CR) and Very Good Partial Response (VGPR)
Percentage of participants with organ response | End of Study (approximately 3 years)
  Organ response for kidney and cardiac is defined as the proportion of baseline organ involved participants who achieve organ response in each corresponding organ. Organ response defined for cardiac: N-terminal brain pronatriuretic peptide (NT-proBNP) response (> 30% and > 300 nanogram per liter [ng/L] decrease in participants with baseline NT-proBNP >= 650 ng/L) or New York Heart Association (NYHA) class response (>= 2 class decrease in participants with baseline NYHA class 3 or 4); for kidney: decrease in proteinuria by >=30% or below 0.5 grams /24 hours without renal progression.
Median hematologic Progression Free Survival (PFS) | End of Study (approximately 3 years)
  Median estimate of months that participants have progression free survival and median estimate is calculated using the Kaplan-Meier methodology
Time to first hematologic response | approximately 12 months
  Measured in months between the date of enrollment and the first efficacy evaluation at which the participant has met the criteria for hematologic complete response.
Time to best hematologic response | approximately 12 months
  Measured in months between the date of enrollment and the best hematologic response the subject achieved while on treatment
Time to hematologic progression | End of Study (approximately 3 years)
  Measured in months between the date of enrollment and the first efficacy evaluation at which the participant has met the criteria for hematologic progression
Duration of hematologic response | End of Study (approximately 3 years)
  Duration of hematologic response is defined as the time between the date of initial documentation of hematologic response (i.e. Complete Response, Very Good Partial Response, Partial Response, No Response and Progressive Disease) to the date of the next hematologic response
Time to next therapy | End of Study (approximately 3 years)
  Measured in months from the date of enrollment to the start date of subsequent treatment for AL amyloidosis
Median organ Progression Free Survival (PFS) | End of Study (approximately 3 years)
  Measured in months between the date of enrollment and the first efficacy evaluation at which the participant has met the criteria for hematologic complete response.
Time to organ response | approximately 12 months
  Measured in months between the date of enrollment and the organ response
Time to organ progression | End of Study (approximately 3 years)
  Measured in months between the date of organ response to organ progression
Duration of organ response | End of Study (approximately 3 years)
  Measured in months between the date of initial documentation of organ response to organ progression

CONTACTS AND LOCATIONS:
Overall Officials: Cara Rosenbaum, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine - Multiple Myeloma Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No